CLINICAL TRIAL: NCT04117711
Title: A Phase 1-2, Dose-Escalating, 4-Part Study to Evaluate the Safety and Pharmacokinetics of Single and Multiple Doses of AT-007 in Healthy Adult Subjects and Adult Subjects With Classic Galactosemia
Brief Title: Safety and Pharmacokinetics of AT-007 in Healthy Subjects and in Adult Subjects With Classic Galactosemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Applied Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AT-007-1001
Record Dates: First submitted 2019-08-23; First posted 2019-10-07 (Actual); Results first posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Classic Galactosemia
Keywords: Classic Galactosemia; Aldose Reductase Inhibition; Galactose, Galactitol
MeSH Terms: conditions — Galactosemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AT-007 (Experimental): AT-007 is a CNS and retina penetrant aldose reductase inhibitor.
  Interventions: Drug: AT-007
- Placebo Comparator (Placebo Comparator): Placebo is used as a comparator to the experimental arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AT-007 — AT-007 will be administered once daily before breakfast. Up to 4 different dose cohorts in part A; up to 4 dose cohorts in part B, up to 2 dose cohorts for part C, and up to 3 dose cohorts for part D will be enrolled in the study. The starting dose in Part A will be 0.5 mg/kg as a single dose. Subsequent doses in Part A and all doses in Parts B, C, and D will be based on the results of previous cohorts and/or previous parts of the study. Part B will start after all subjects in Part A have completed the study. Cohort C1 will be conducted simultaneously with Cohort B3 and using the same dose as Cohort B2. The dose for Cohort D1 will not be higher than the dose for Cohort B2. The second and third cohorts in Part D (D2 and D3) will not start until after all subjects in Cohorts B3 and B4, respectively, have completed the study and the dose levels will not be higher than those for Cohorts B3 and B4, respectively.
  Other Names: Govorestat
  Arms: AT-007
Drug: Placebo — Matching placebo will be administered once in the morning before breakfast
  Arms: Placebo Comparator

SUMMARY:
This study is a first-in-human, randomized, placebo-controlled, 4-Part, single ascending dose (SAD) and multiple ascending dose (MAD) study in healthy adult subjects and adult subjects with Classic Galactosemia.

DETAILED DESCRIPTION:
The study is designed to assess the safety and PK of AT-007 in healthy subjects and subjects with Classic Galactosemia as well as the effect of AT-007 on biomarkers of galactose metabolism (galactose, galactitol, and other galactose metabolites) in subjects with Classic Galactosemia.

This study consists of 4 parts:

* Part A (SAD) in 32 healthy subjects. Once daily oral escalating dose (6 active, 2 placebo).
* Part B and C (MAD for 7 days) in 36 healthy subjects. Once daily multiple daily dosing (8 active, 2 placebo per each dose cohort).
* Part D (SAD followed by MAD for 27 days) in 18 subjects with Classic Galactosemia. Once daily followed by multiple daily oral dosing (6 active, 2 placebo for each dose cohort).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Classic Galactosemia confirmed by evidence of absent or significantly decreased (<1%) GALT activity in red blood cells and by GALT gene analysis
* Urine galactitol >100 mmol/mol creatinine
* Galactose-restricted diet

Exclusion Criteria:

* Complications of CG resulting in disability that, in the opinion of the Investigator, may prevent the subject from completing all study requirements (e.g., severe neurological deficits, severe cognitive impairment, or severe language difficulty).
* Renal disease (eGFR < 90 mL/min/1.73 m2 or albuminuria).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2019-06-21 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2021-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Green, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (4):
- United States (4):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Brigham and Women's Hospital, Boston, Massachusetts
  - ICON Clinical Research, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A Cohort 1: AT-007 0.5mg/kg; Part A Cohort 2: AT-007 5mg/kg; Part A Cohort 3: AT-007 10mg/kg; Part A Cohort 4: AT-007 20mg/kg; Part A Cohort 5: AT-007 40mg/kg: AT-007 administered once daily before breakfast as a single dose.
- Part A: Placebo Comparator: Placebo: Matching placebo will be administered once in the morning before breakfast as a single dose
- Part B & C: AT-007 5mg/kg; Part B & C: AT-007 10mg/kg; Part B & C: AT-007 20mg/kg; Part B & C: AT-007 40mg/kg; Part B &C: Placebo Comparator: Part B and Part C are combined with results pooled for each dose level. Healthy adult volunteers received multiple doses of AT-007 once daily for 7 days.
- Part D Cohort 1: AT-007 5mg/kg; Part D Cohort 2: AT-007 20mg/kg; Part D Cohort 3: AT-007 40mg/kg: AT-007 administered as a single dose once followed by a 5-day wash followed by 28 days of dosing.
- Part D Cohort 1 (Placebo) Then Cohort 2 (AT-007 20mg/kg: Placebo administered as a single dose once followed by a 5-day wash followed by 28 days of dosing in Cohort 1. Then, after washout, AT-007 administered as a single dose once followed by a 5-day wash followed by 28 days of dosing in Cohort 2.
- Part D Cohort 1 (AT-007 5mg/kg) Then Cohort 3 (AT-007 40mg/kg): AT-007 administered as a single dose once followed by a 5-day wash followed by 28 days of dosing for each dosing cohort after a washout between cohort dosing.
- Part D Cohort 1 (Placebo) Then Cohort 3 (AT-007 40mg/kg): Placebo administered as a single dose once followed by a 5-day wash followed by 28 days of dosing in Cohort 1. After washout, AT-007 administered as a single dose once followed by a 5-day wash followed by 28 days of dosing in Cohort 3.
- Part D Cohort 2 (AT-007 20mg/kg) Then Cohort 3 (AT-007 40mg/kg): AT-007 administered as a single dose once followed by a 5-day wash followed by 28 days of dosing for each cohort with washout between cohorts.
- Part D: Placebo Comparator: Placebo administered as a single dose once followed by a 5-day wash followed by 28 days of dosing.
- Part D Extension Cohort 1: AT-007 20mg/kg; Part D Extension Cohort 2: 40mg/kg: Adults with Classic Galactosemia, daily doses of AT-007 for 90 days
- Part D Extension: Placebo Compartor: Adults with Classic Galactosemia, daily doses of placebo for 90 days
Period: Part A Cohort 1
Arm/Group | Part A Cohort 1: AT-007 0.5mg/kg | Part A Cohort 2: AT-007 5mg/kg | Part A Cohort 3: AT-007 10mg/kg | Part A Cohort 4: AT-007 20mg/kg | Part A Cohort 5: AT-007 40mg/kg | Part A: Placebo Comparator | Part B & C: AT-007 5mg/kg | Part B & C: AT-007 10mg/kg | Part B & C: AT-007 20mg/kg | Part B & C: AT-007 40mg/kg | Part B &C: Placebo Comparator | Part D Cohort 1: AT-007 5mg/kg | Part D Cohort 1 (Placebo) Then Cohort 2 (AT-007 20mg/kg | Part D Cohort 1 (AT-007 5mg/kg) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 1 (Placebo) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 2: AT-007 20mg/kg | Part D Cohort 2 (AT-007 20mg/kg) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 3: AT-007 40mg/kg | Part D: Placebo Comparator | Part D Extension Cohort 1: AT-007 20mg/kg | Part D Extension Cohort 2: 40mg/kg | Part D Extension: Placebo Compartor
Started | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A Cohort 2
Arm/Group | Part A Cohort 1: AT-007 0.5mg/kg | Part A Cohort 2: AT-007 5mg/kg | Part A Cohort 3: AT-007 10mg/kg | Part A Cohort 4: AT-007 20mg/kg | Part A Cohort 5: AT-007 40mg/kg | Part A: Placebo Comparator | Part B & C: AT-007 5mg/kg | Part B & C: AT-007 10mg/kg | Part B & C: AT-007 20mg/kg | Part B & C: AT-007 40mg/kg | Part B &C: Placebo Comparator | Part D Cohort 1: AT-007 5mg/kg | Part D Cohort 1 (Placebo) Then Cohort 2 (AT-007 20mg/kg | Part D Cohort 1 (AT-007 5mg/kg) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 1 (Placebo) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 2: AT-007 20mg/kg | Part D Cohort 2 (AT-007 20mg/kg) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 3: AT-007 40mg/kg | Part D: Placebo Comparator | Part D Extension Cohort 1: AT-007 20mg/kg | Part D Extension Cohort 2: 40mg/kg | Part D Extension: Placebo Compartor
Started | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A Cohort 3
Arm/Group | Part A Cohort 1: AT-007 0.5mg/kg | Part A Cohort 2: AT-007 5mg/kg | Part A Cohort 3: AT-007 10mg/kg | Part A Cohort 4: AT-007 20mg/kg | Part A Cohort 5: AT-007 40mg/kg | Part A: Placebo Comparator | Part B & C: AT-007 5mg/kg | Part B & C: AT-007 10mg/kg | Part B & C: AT-007 20mg/kg | Part B & C: AT-007 40mg/kg | Part B &C: Placebo Comparator | Part D Cohort 1: AT-007 5mg/kg | Part D Cohort 1 (Placebo) Then Cohort 2 (AT-007 20mg/kg | Part D Cohort 1 (AT-007 5mg/kg) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 1 (Placebo) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 2: AT-007 20mg/kg | Part D Cohort 2 (AT-007 20mg/kg) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 3: AT-007 40mg/kg | Part D: Placebo Comparator | Part D Extension Cohort 1: AT-007 20mg/kg | Part D Extension Cohort 2: 40mg/kg | Part D Extension: Placebo Compartor
Started | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A Cohort 4
Arm/Group | Part A Cohort 1: AT-007 0.5mg/kg | Part A Cohort 2: AT-007 5mg/kg | Part A Cohort 3: AT-007 10mg/kg | Part A Cohort 4: AT-007 20mg/kg | Part A Cohort 5: AT-007 40mg/kg | Part A: Placebo Comparator | Part B & C: AT-007 5mg/kg | Part B & C: AT-007 10mg/kg | Part B & C: AT-007 20mg/kg | Part B & C: AT-007 40mg/kg | Part B &C: Placebo Comparator | Part D Cohort 1: AT-007 5mg/kg | Part D Cohort 1 (Placebo) Then Cohort 2 (AT-007 20mg/kg | Part D Cohort 1 (AT-007 5mg/kg) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 1 (Placebo) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 2: AT-007 20mg/kg | Part D Cohort 2 (AT-007 20mg/kg) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 3: AT-007 40mg/kg | Part D: Placebo Comparator | Part D Extension Cohort 1: AT-007 20mg/kg | Part D Extension Cohort 2: 40mg/kg | Part D Extension: Placebo Compartor
Started | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A Cohort 5
Arm/Group | Part A Cohort 1: AT-007 0.5mg/kg | Part A Cohort 2: AT-007 5mg/kg | Part A Cohort 3: AT-007 10mg/kg | Part A Cohort 4: AT-007 20mg/kg | Part A Cohort 5: AT-007 40mg/kg | Part A: Placebo Comparator | Part B & C: AT-007 5mg/kg | Part B & C: AT-007 10mg/kg | Part B & C: AT-007 20mg/kg | Part B & C: AT-007 40mg/kg | Part B &C: Placebo Comparator | Part D Cohort 1: AT-007 5mg/kg | Part D Cohort 1 (Placebo) Then Cohort 2 (AT-007 20mg/kg | Part D Cohort 1 (AT-007 5mg/kg) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 1 (Placebo) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 2: AT-007 20mg/kg | Part D Cohort 2 (AT-007 20mg/kg) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 3: AT-007 40mg/kg | Part D: Placebo Comparator | Part D Extension Cohort 1: AT-007 20mg/kg | Part D Extension Cohort 2: 40mg/kg | Part D Extension: Placebo Compartor
Started | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A Placebo Comparator
Arm/Group | Part A Cohort 1: AT-007 0.5mg/kg | Part A Cohort 2: AT-007 5mg/kg | Part A Cohort 3: AT-007 10mg/kg | Part A Cohort 4: AT-007 20mg/kg | Part A Cohort 5: AT-007 40mg/kg | Part A: Placebo Comparator | Part B & C: AT-007 5mg/kg | Part B & C: AT-007 10mg/kg | Part B & C: AT-007 20mg/kg | Part B & C: AT-007 40mg/kg | Part B &C: Placebo Comparator | Part D Cohort 1: AT-007 5mg/kg | Part D Cohort 1 (Placebo) Then Cohort 2 (AT-007 20mg/kg | Part D Cohort 1 (AT-007 5mg/kg) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 1 (Placebo) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 2: AT-007 20mg/kg | Part D Cohort 2 (AT-007 20mg/kg) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 3: AT-007 40mg/kg | Part D: Placebo Comparator | Part D Extension Cohort 1: AT-007 20mg/kg | Part D Extension Cohort 2: 40mg/kg | Part D Extension: Placebo Compartor
Started | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B & C AT-007 5mg/kg Cohort
Arm/Group | Part A Cohort 1: AT-007 0.5mg/kg | Part A Cohort 2: AT-007 5mg/kg | Part A Cohort 3: AT-007 10mg/kg | Part A Cohort 4: AT-007 20mg/kg | Part A Cohort 5: AT-007 40mg/kg | Part A: Placebo Comparator | Part B & C: AT-007 5mg/kg | Part B & C: AT-007 10mg/kg | Part B & C: AT-007 20mg/kg | Part B & C: AT-007 40mg/kg | Part B &C: Placebo Comparator | Part D Cohort 1: AT-007 5mg/kg | Part D Cohort 1 (Placebo) Then Cohort 2 (AT-007 20mg/kg | Part D Cohort 1 (AT-007 5mg/kg) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 1 (Placebo) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 2: AT-007 20mg/kg | Part D Cohort 2 (AT-007 20mg/kg) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 3: AT-007 40mg/kg | Part D: Placebo Comparator | Part D Extension Cohort 1: AT-007 20mg/kg | Part D Extension Cohort 2: 40mg/kg | Part D Extension: Placebo Compartor
Started | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B & C AT-007 10mg/kg Cohort
Arm/Group | Part A Cohort 1: AT-007 0.5mg/kg | Part A Cohort 2: AT-007 5mg/kg | Part A Cohort 3: AT-007 10mg/kg | Part A Cohort 4: AT-007 20mg/kg | Part A Cohort 5: AT-007 40mg/kg | Part A: Placebo Comparator | Part B & C: AT-007 5mg/kg | Part B & C: AT-007 10mg/kg | Part B & C: AT-007 20mg/kg | Part B & C: AT-007 40mg/kg | Part B &C: Placebo Comparator | Part D Cohort 1: AT-007 5mg/kg | Part D Cohort 1 (Placebo) Then Cohort 2 (AT-007 20mg/kg | Part D Cohort 1 (AT-007 5mg/kg) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 1 (Placebo) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 2: AT-007 20mg/kg | Part D Cohort 2 (AT-007 20mg/kg) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 3: AT-007 40mg/kg | Part D: Placebo Comparator | Part D Extension Cohort 1: AT-007 20mg/kg | Part D Extension Cohort 2: 40mg/kg | Part D Extension: Placebo Compartor
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B & C AT-007 20mg/kg Cohort
Arm/Group | Part A Cohort 1: AT-007 0.5mg/kg | Part A Cohort 2: AT-007 5mg/kg | Part A Cohort 3: AT-007 10mg/kg | Part A Cohort 4: AT-007 20mg/kg | Part A Cohort 5: AT-007 40mg/kg | Part A: Placebo Comparator | Part B & C: AT-007 5mg/kg | Part B & C: AT-007 10mg/kg | Part B & C: AT-007 20mg/kg | Part B & C: AT-007 40mg/kg | Part B &C: Placebo Comparator | Part D Cohort 1: AT-007 5mg/kg | Part D Cohort 1 (Placebo) Then Cohort 2 (AT-007 20mg/kg | Part D Cohort 1 (AT-007 5mg/kg) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 1 (Placebo) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 2: AT-007 20mg/kg | Part D Cohort 2 (AT-007 20mg/kg) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 3: AT-007 40mg/kg | Part D: Placebo Comparator | Part D Extension Cohort 1: AT-007 20mg/kg | Part D Extension Cohort 2: 40mg/kg | Part D Extension: Placebo Compartor
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B & C AT-007 40mg/kg
Arm/Group | Part A Cohort 1: AT-007 0.5mg/kg | Part A Cohort 2: AT-007 5mg/kg | Part A Cohort 3: AT-007 10mg/kg | Part A Cohort 4: AT-007 20mg/kg | Part A Cohort 5: AT-007 40mg/kg | Part A: Placebo Comparator | Part B & C: AT-007 5mg/kg | Part B & C: AT-007 10mg/kg | Part B & C: AT-007 20mg/kg | Part B & C: AT-007 40mg/kg | Part B &C: Placebo Comparator | Part D Cohort 1: AT-007 5mg/kg | Part D Cohort 1 (Placebo) Then Cohort 2 (AT-007 20mg/kg | Part D Cohort 1 (AT-007 5mg/kg) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 1 (Placebo) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 2: AT-007 20mg/kg | Part D Cohort 2 (AT-007 20mg/kg) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 3: AT-007 40mg/kg | Part D: Placebo Comparator | Part D Extension Cohort 1: AT-007 20mg/kg | Part D Extension Cohort 2: 40mg/kg | Part D Extension: Placebo Compartor
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B & C Placebo Comparator
Arm/Group | Part A Cohort 1: AT-007 0.5mg/kg | Part A Cohort 2: AT-007 5mg/kg | Part A Cohort 3: AT-007 10mg/kg | Part A Cohort 4: AT-007 20mg/kg | Part A Cohort 5: AT-007 40mg/kg | Part A: Placebo Comparator | Part B & C: AT-007 5mg/kg | Part B & C: AT-007 10mg/kg | Part B & C: AT-007 20mg/kg | Part B & C: AT-007 40mg/kg | Part B &C: Placebo Comparator | Part D Cohort 1: AT-007 5mg/kg | Part D Cohort 1 (Placebo) Then Cohort 2 (AT-007 20mg/kg | Part D Cohort 1 (AT-007 5mg/kg) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 1 (Placebo) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 2: AT-007 20mg/kg | Part D Cohort 2 (AT-007 20mg/kg) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 3: AT-007 40mg/kg | Part D: Placebo Comparator | Part D Extension Cohort 1: AT-007 20mg/kg | Part D Extension Cohort 2: 40mg/kg | Part D Extension: Placebo Compartor
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part D Cohort 1
Arm/Group | Part A Cohort 1: AT-007 0.5mg/kg | Part A Cohort 2: AT-007 5mg/kg | Part A Cohort 3: AT-007 10mg/kg | Part A Cohort 4: AT-007 20mg/kg | Part A Cohort 5: AT-007 40mg/kg | Part A: Placebo Comparator | Part B & C: AT-007 5mg/kg | Part B & C: AT-007 10mg/kg | Part B & C: AT-007 20mg/kg | Part B & C: AT-007 40mg/kg | Part B &C: Placebo Comparator | Part D Cohort 1: AT-007 5mg/kg | Part D Cohort 1 (Placebo) Then Cohort 2 (AT-007 20mg/kg | Part D Cohort 1 (AT-007 5mg/kg) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 1 (Placebo) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 2: AT-007 20mg/kg | Part D Cohort 2 (AT-007 20mg/kg) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 3: AT-007 40mg/kg | Part D: Placebo Comparator | Part D Extension Cohort 1: AT-007 20mg/kg | Part D Extension Cohort 2: 40mg/kg | Part D Extension: Placebo Compartor
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part D Cohort 2
Arm/Group | Part A Cohort 1: AT-007 0.5mg/kg | Part A Cohort 2: AT-007 5mg/kg | Part A Cohort 3: AT-007 10mg/kg | Part A Cohort 4: AT-007 20mg/kg | Part A Cohort 5: AT-007 40mg/kg | Part A: Placebo Comparator | Part B & C: AT-007 5mg/kg | Part B & C: AT-007 10mg/kg | Part B & C: AT-007 20mg/kg | Part B & C: AT-007 40mg/kg | Part B &C: Placebo Comparator | Part D Cohort 1: AT-007 5mg/kg | Part D Cohort 1 (Placebo) Then Cohort 2 (AT-007 20mg/kg | Part D Cohort 1 (AT-007 5mg/kg) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 1 (Placebo) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 2: AT-007 20mg/kg | Part D Cohort 2 (AT-007 20mg/kg) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 3: AT-007 40mg/kg | Part D: Placebo Comparator | Part D Extension Cohort 1: AT-007 20mg/kg | Part D Extension Cohort 2: 40mg/kg | Part D Extension: Placebo Compartor
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part D Cohort 3
Arm/Group | Part A Cohort 1: AT-007 0.5mg/kg | Part A Cohort 2: AT-007 5mg/kg | Part A Cohort 3: AT-007 10mg/kg | Part A Cohort 4: AT-007 20mg/kg | Part A Cohort 5: AT-007 40mg/kg | Part A: Placebo Comparator | Part B & C: AT-007 5mg/kg | Part B & C: AT-007 10mg/kg | Part B & C: AT-007 20mg/kg | Part B & C: AT-007 40mg/kg | Part B &C: Placebo Comparator | Part D Cohort 1: AT-007 5mg/kg | Part D Cohort 1 (Placebo) Then Cohort 2 (AT-007 20mg/kg | Part D Cohort 1 (AT-007 5mg/kg) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 1 (Placebo) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 2: AT-007 20mg/kg | Part D Cohort 2 (AT-007 20mg/kg) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 3: AT-007 40mg/kg | Part D: Placebo Comparator | Part D Extension Cohort 1: AT-007 20mg/kg | Part D Extension Cohort 2: 40mg/kg | Part D Extension: Placebo Compartor
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part D Placebo Comparator
Arm/Group | Part A Cohort 1: AT-007 0.5mg/kg | Part A Cohort 2: AT-007 5mg/kg | Part A Cohort 3: AT-007 10mg/kg | Part A Cohort 4: AT-007 20mg/kg | Part A Cohort 5: AT-007 40mg/kg | Part A: Placebo Comparator | Part B & C: AT-007 5mg/kg | Part B & C: AT-007 10mg/kg | Part B & C: AT-007 20mg/kg | Part B & C: AT-007 40mg/kg | Part B &C: Placebo Comparator | Part D Cohort 1: AT-007 5mg/kg | Part D Cohort 1 (Placebo) Then Cohort 2 (AT-007 20mg/kg | Part D Cohort 1 (AT-007 5mg/kg) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 1 (Placebo) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 2: AT-007 20mg/kg | Part D Cohort 2 (AT-007 20mg/kg) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 3: AT-007 40mg/kg | Part D: Placebo Comparator | Part D Extension Cohort 1: AT-007 20mg/kg | Part D Extension Cohort 2: 40mg/kg | Part D Extension: Placebo Compartor
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part D Extension Cohort 1
Arm/Group | Part A Cohort 1: AT-007 0.5mg/kg | Part A Cohort 2: AT-007 5mg/kg | Part A Cohort 3: AT-007 10mg/kg | Part A Cohort 4: AT-007 20mg/kg | Part A Cohort 5: AT-007 40mg/kg | Part A: Placebo Comparator | Part B & C: AT-007 5mg/kg | Part B & C: AT-007 10mg/kg | Part B & C: AT-007 20mg/kg | Part B & C: AT-007 40mg/kg | Part B &C: Placebo Comparator | Part D Cohort 1: AT-007 5mg/kg | Part D Cohort 1 (Placebo) Then Cohort 2 (AT-007 20mg/kg | Part D Cohort 1 (AT-007 5mg/kg) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 1 (Placebo) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 2: AT-007 20mg/kg | Part D Cohort 2 (AT-007 20mg/kg) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 3: AT-007 40mg/kg | Part D: Placebo Comparator | Part D Extension Cohort 1: AT-007 20mg/kg | Part D Extension Cohort 2: 40mg/kg | Part D Extension: Placebo Compartor
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Period: Part D Extension Cohort 2
Arm/Group | Part A Cohort 1: AT-007 0.5mg/kg | Part A Cohort 2: AT-007 5mg/kg | Part A Cohort 3: AT-007 10mg/kg | Part A Cohort 4: AT-007 20mg/kg | Part A Cohort 5: AT-007 40mg/kg | Part A: Placebo Comparator | Part B & C: AT-007 5mg/kg | Part B & C: AT-007 10mg/kg | Part B & C: AT-007 20mg/kg | Part B & C: AT-007 40mg/kg | Part B &C: Placebo Comparator | Part D Cohort 1: AT-007 5mg/kg | Part D Cohort 1 (Placebo) Then Cohort 2 (AT-007 20mg/kg | Part D Cohort 1 (AT-007 5mg/kg) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 1 (Placebo) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 2: AT-007 20mg/kg | Part D Cohort 2 (AT-007 20mg/kg) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 3: AT-007 40mg/kg | Part D: Placebo Comparator | Part D Extension Cohort 1: AT-007 20mg/kg | Part D Extension Cohort 2: 40mg/kg | Part D Extension: Placebo Compartor
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Period: Part D Extension Placebo Comparator
Arm/Group | Part A Cohort 1: AT-007 0.5mg/kg | Part A Cohort 2: AT-007 5mg/kg | Part A Cohort 3: AT-007 10mg/kg | Part A Cohort 4: AT-007 20mg/kg | Part A Cohort 5: AT-007 40mg/kg | Part A: Placebo Comparator | Part B & C: AT-007 5mg/kg | Part B & C: AT-007 10mg/kg | Part B & C: AT-007 20mg/kg | Part B & C: AT-007 40mg/kg | Part B &C: Placebo Comparator | Part D Cohort 1: AT-007 5mg/kg | Part D Cohort 1 (Placebo) Then Cohort 2 (AT-007 20mg/kg | Part D Cohort 1 (AT-007 5mg/kg) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 1 (Placebo) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 2: AT-007 20mg/kg | Part D Cohort 2 (AT-007 20mg/kg) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 3: AT-007 40mg/kg | Part D: Placebo Comparator | Part D Extension Cohort 1: AT-007 20mg/kg | Part D Extension Cohort 2: 40mg/kg | Part D Extension: Placebo Compartor
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Part A Cohort 1: AT-007 0.5mg/kg; Part A Cohort 2: AT-007 5mg/kg; Part A Cohort 3: AT-007 10mg/kg; Part A Cohort 4: AT-007 20mg/kg; Part A Cohort 5: AT-007 40mg/kg; Part A Placebo Comparator: Baseline characteristics of the healthy adult subjects enrolled in Part A were well-balanced between active and placebo across all dosing cohorts.
- Part B & C AT-007 5mg/kg Cohort; Part B & C AT-007 10mg/kg Cohort; Part B & C AT-007 20mg/kg Cohort; Part B & C AT-007 40mg/kg Cohort; Part B & C Placebo Comparator: Baseline characteristics of the healthy adult subjects enrolled in Part B & C were well-balanced between active and placebo across all dosing cohorts.
- Part D Cohort 1: AT-007 5mg/kg; Part D Cohort 1 (Placebo) Then Cohort 2 (AT-007 20mg/kg); Part D Cohort 1 (AT-007 5mg/kg) Then Cohort 3 (AT-007 40mg/kg); Part D Cohort 1 (Placebo) Then Cohort 3 (AT-007 40mg/kg); Part D Cohort 2: AT-007 20mg/kg; Part D Cohort 2 (AT-007 20mg/kg) Then Chort 3 (AT-007 40mg/kg); Part D Cohort 3: AT-007 40mg/kg; Part D Placebo Comparator: Baseline characteristics of the adult subjects with Classic Galactosemia enrolled in Part D were well-balanced between active and placebo across all dosing cohorts.
- Part D Extension Placebo Comparator; Part D Extension Cohort 1: AT-007 20mg/kg; Part D Extension Cohort 2: AT-007 40mg/kg: Baseline characteristics of the adult subjects with Classic Galactosemia enrolled in Part D Extension were well-balanced between active and placebo across all dosing cohorts.
- Total: Total of all reporting groups
Arm/Group | Part A Cohort 1: AT-007 0.5mg/kg | Part A Cohort 2: AT-007 5mg/kg | Part A Cohort 3: AT-007 10mg/kg | Part A Cohort 4: AT-007 20mg/kg | Part A Cohort 5: AT-007 40mg/kg | Part A Placebo Comparator | Part B & C AT-007 5mg/kg Cohort | Part B & C AT-007 10mg/kg Cohort | Part B & C AT-007 20mg/kg Cohort | Part B & C AT-007 40mg/kg Cohort | Part B & C Placebo Comparator | Part D Cohort 1: AT-007 5mg/kg | Part D Cohort 1 (Placebo) Then Cohort 2 (AT-007 20mg/kg) | Part D Cohort 1 (AT-007 5mg/kg) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 1 (Placebo) Then Cohort 3 (AT-007 40mg/kg) | Part D Cohort 2: AT-007 20mg/kg | Part D Cohort 2 (AT-007 20mg/kg) Then Chort 3 (AT-007 40mg/kg) | Part D Cohort 3: AT-007 40mg/kg | Part D Placebo Comparator | Part D Extension Placebo Comparator | Part D Extension Cohort 1: AT-007 20mg/kg | Part D Extension Cohort 2: AT-007 40mg/kg | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10 | 6 | 8 | 10 | 9 | 8 | 3 | 1 | 1 | 1 | 2 | 1 | 1 | 4 | 4 | 9 | 2 | 110
Age, Continuous [Median (Full Range); unit: years] | 42.5 [37 to 49] | 54.0 [47 to 58] | 35.0 [27 to 45] | 44.0 [39 to 52] | 31.5 [25 to 43] | 54.5 [39 to 64] | 32.5 [29 to 53] | 35.5 [30 to 40] | 35.0 [28 to 37] | 27.0 [23 to 37] | 37 [33 to 41.5] | 19.5 [18 to 21] | 37 [37 to 37] | 50 [50 to 50] | 19 [19 to 19] | 20.5 [19 to 22] | 28 [28 to 28] | 43 [43 to 43] | 32 [23 to 44] | 29.5 [20 to 41] | 22.0 [19 to 25] | 36.0 [22 to 50] | NA [NA to NA] — As per the SAP, healthy adults cannot be combined with the disease population.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 2 | 4 | 4 | 8 | 5 | 3 | 4 | 5 | 3 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 3 | 3 | 0 | 56
  Male | 4 | 1 | 4 | 2 | 2 | 2 | 1 | 5 | 6 | 4 | 5 | 2 | 1 | 1 | 0 | 1 | 1 | 1 | 2 | 1 | 6 | 2 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 2 | 2 | 3 | 9 | 4 | 3 | 6 | 5 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 43
  Not Hispanic or Latino | 5 | 1 | 4 | 4 | 3 | 1 | 2 | 5 | 4 | 4 | 5 | 3 | 1 | 1 | 1 | 2 | 1 | 1 | 4 | 4 | 9 | 2 | 67
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Asian | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 2 | 3 | 2 | 1 | 1 | 4 | 3 | 2 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 24
  White | 4 | 6 | 3 | 3 | 3 | 9 | 5 | 4 | 6 | 7 | 3 | 3 | 1 | 1 | 1 | 2 | 1 | 1 | 4 | 4 | 9 | 2 | 82
  More than one race | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 6 | 6 | 10 | 6 | 8 | 10 | 9 | 8 | 3 | 1 | 1 | 1 | 2 | 1 | 1 | 4 | 4 | 9 | 2 | 110
Galactitol [Median (Full Range); unit: ng/mL] — Galactitol is a disease specific pharmakodynamic marker in Classic Galactosemia and therefore was only collected and measured in Part D and Part D Extension. Galactitol is NOT measurable in healthy people because they do not produce it; as such and as per protocol it was not collected and not measured in healthy adults. This means that no healthy adults had galactitol measured so it is not present for Part A, Part B, or Part C. The units are ng/mL and it's measured in plasma. Population: Galactitol is NOT measurable in healthy people because they do not produce it; as such and as per protocol it was not collected and not measured in healthy adults. This means that no healthy adults had galactitol measured so it is not present for Part A, Part B, or Part C.
  ng/mL
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 1 | 2 | 1 | 1 | 4 | 4 | 9 | 2 | 29
    (all) |  |  |  |  |  |  |  |  |  |  |  | 2490 [2200 to 2580] | 2380 [2380 to 2380] | 2140 [2140 to 2140] | 2360 [2360 to 2360] | 2170 [2060 to 2280] | 2340 [2340 to 2340] | 2810 [2810 to 2810] | 2480 [1995 to 3420] | 2612.5 [1960 to 3670] | 2300 [1780 to 2775] | NA [NA to NA] — As was evaluated by the DMC and directed by their independent review, if the 20 mg/kg and 40 mg/kg doses resulted in equivalent galactitol reduction, Part D Extension Cohort 2 40mg/kg would be stopped early. This was true and Part D Extension was stopped at at Day 30 and no further data was collected. | 2434.4 [1950 to 3670]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: To evaluate the safety and tolerability of AT-007 after administration to healthy subjects, including clinically-significant changes in clinical laboratory test results, physical examination findings, vital sign evaluations, and electrocardiogram results.
Time Frame: Events after 1 day of administration.
Population: All subjects dosed were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Part A Cohort 1: AT-007 0.5mg/kg; Part A Cohort 2: AT-007 5mg/kg; Part A Cohort 3: AT-007 10mg/kg; Part A Cohort 4: AT-007 20mg/kg; Part A Cohort 5: AT-007 40mg/kg: Single doses of orally administered AT-007 were administered to Healthy Adult Subjects and all TEAEs recorded.
- Part A: Placebo Comparator: Single doses of orally administered matched-placebo were administered to Healthy Adult Subjects and all TEAEs recorded.
Arm/Group | Part A Cohort 1: AT-007 0.5mg/kg | Part A Cohort 2: AT-007 5mg/kg | Part A Cohort 3: AT-007 10mg/kg | Part A Cohort 4: AT-007 20mg/kg | Part A Cohort 5: AT-007 40mg/kg | Part A: Placebo Comparator
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10
Participants | 1 | 0 | 0 | 2 | 1 | 2

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: To evaluate the safety and tolerability of AT-007 after multiple ascending doses are administered to healthy subjects, including clinically-significant changes in clinical laboratory test results, physical examination findings, vital sign evaluations, and electrocardiogram results. Part B and Part C are combined.
Time Frame: 7 Days after Dosing
Population: All subjects dosed were analyzed
Measure: Count of Participants; unit: Participants
Groups:
- Part B & C AT-007 5mg/kg Cohort; Part B & C AT-007 10mg/kg Cohort; Part B & C AT-007 20mg/kg Cohort; Part B & C AT-007 40mg/kg Cohort: Multiple doses of orally administered AT-007 were administered to healthy adult subjects and all TEAEs recorded.
- Part B & C Placebo Comparator: Multiple doses of orally administered matched-placebo were administered to healthy adult subjects and all TEAEs recorded.
Arm/Group | Part B & C AT-007 5mg/kg Cohort | Part B & C AT-007 10mg/kg Cohort | Part B & C AT-007 20mg/kg Cohort | Part B & C AT-007 40mg/kg Cohort | Part B & C Placebo Comparator
Number analyzed (Participants) | 6 | 8 | 10 | 9 | 8
Participants | 1 | 2 | 3 | 1 | 2

3. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: To evaluate the safety and tolerability of AT-007 after multiple doses administered to Classic Galactosemia Patients, including clinically-significant changes in clinical laboratory test results, physical examination findings, vital sign evaluations, and electrocardiogram results.
Time Frame: 28 Days of Dosing
Population: All subjects dosed were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Part D Cohort 1: AT-007 5mg/kg; Part D Cohort 2: AT-007 20mg/kg; Part D Cohort 3: AT-007 40mg/kg: Multiple doses of orally administered AT-007 were administered to adult subjects with Classic Galactosemia and all TEAEs were recorded.
- Part D Placebo Comparator: Multiple doses of orally administered matched placebo were administered to adult subjects with Classic Galactosemia and all TEAEs were recorded.
Arm/Group | Part D Cohort 1: AT-007 5mg/kg | Part D Cohort 2: AT-007 20mg/kg | Part D Cohort 3: AT-007 40mg/kg | Part D Placebo Comparator
Number analyzed (Participants) | 4 | 4 | 4 | 6
Participants | 3 | 1 | 2 | 2

4. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: To evaluate the safety and tolerability of AT-007 administered to Classic Galactosemia Patients, including clinically-significant changes in clinical laboratory test results, physical examination findings, vital sign evaluations, and electrocardiogram results.
Time Frame: 90 Days after Dosing
Population: All subjects dosed were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Part D Extension Cohort 1: AT-007 20mg/kg; Part D Extension Cohort 2: AT-007 40mg/kg: Multiple doses of AT-007 were orally administered to adult subjects with Classic Galactosemia and all TEAEs were recorded.
- Part D Extension Placebo Comparator: Multiple doses of matched-placebo were orally administered to adult subjects with Classic Galactosemia and all TEAEs were recorded.
Arm/Group | Part D Extension Cohort 1: AT-007 20mg/kg | Part D Extension Cohort 2: AT-007 40mg/kg | Part D Extension Placebo Comparator
Number analyzed (Participants) | 9 | 2 | 4
Participants | 7 | 1 | 2

5. Secondary Outcome: Cmax of AT-007
Description: Maximum (peak) plasma drug concentration
Time Frame: Part A: Sampling- predose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 36, 48 hrs Parts B, C, D: Day of Last Dose for each Part- predose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 36, 48 hrs D Extension: Day 30, 60, 90- predose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 36, 48 hrs
Population: Part D Extension Cohort 2 40mg/kg ended early at Day 30 as recommended by Monitoring Committee. As such, only 1 subject has D30 data available; the other subject did not have enough blood samples to calculate.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/mL
Groups:
- Part A Cohort 1: AT-007 0.5mg/kg; Part A Cohort 2: AT-007 5mg/kg; Part A Cohort 3: AT-007 10mg/kg; Part A Cohort 4: AT-007 20mg/kg; Part A Cohort 5: AT-007 40mg/kg: Following a single dose of AT-007 to Healthy Adult Subjects, sequential sampling was performed and Cmax calculated.
- Part B & C Cohort 1: AT-007 5mg/kg; Part B & C Cohort 2: AT-007 10mg/kg; Part B & C Cohort 3: AT-007 20mg/kg; Part B & C Cohort 4: AT-007 40mg/kg: Following multiple QD dose administration of AT-007 for 7 days in Healthy Adult Subjects, Cmax was calculated. Day 7 is presented as it reflects steady state.
- Part D Cohort 1: AT-007 5mg/kg; Part D Cohort 2: AT-007 20mg/kg; Part D Cohort 3: AT-007 40mg/kg: Following multiple QD dose administration of AT-007 in Adults with Classic Galactosemia, Cmax was calculated. Day 32 is presented as it reflects steady state.
- Part D Extension Cohort 1: AT-007 20mg/kg DAY 30; Part D Extension Cohort 1: AT-007 20mg/kg DAY 60; Part D Extension Cohort 1: AT-007 20mg/kg DAY 90: Following multiple QD dose administration of AT-007 in Adults with Classic Galactosemia, Cmax was calculated. Days 30, 60, and 90 are presented to reflect values over time.
- Part D Extension Cohort 2: AT-007 40mg/kg DAY 30: Following multiple QD dose administration of AT-007 in Adults with Classic Galactosemia
Arm/Group | Part A Cohort 1: AT-007 0.5mg/kg | Part A Cohort 2: AT-007 5mg/kg | Part A Cohort 3: AT-007 10mg/kg | Part A Cohort 4: AT-007 20mg/kg | Part A Cohort 5: AT-007 40mg/kg | Part B & C Cohort 1: AT-007 5mg/kg | Part B & C Cohort 2: AT-007 10mg/kg | Part B & C Cohort 3: AT-007 20mg/kg | Part B & C Cohort 4: AT-007 40mg/kg | Part D Cohort 1: AT-007 5mg/kg | Part D Cohort 2: AT-007 20mg/kg | Part D Cohort 3: AT-007 40mg/kg | Part D Extension Cohort 1: AT-007 20mg/kg DAY 30 | Part D Extension Cohort 1: AT-007 20mg/kg DAY 60 | Part D Extension Cohort 1: AT-007 20mg/kg DAY 90 | Part D Extension Cohort 2: AT-007 40mg/kg DAY 30
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 9 | 7 | 4 | 4 | 4 | 9 | 8 | 6 | 1
microgram/mL | 1.53 (55.2) | 8.92 (31.4) | 15.2 (49.5) | 27 (103) | 57.4 (23.2) | 15.2 (45.0) | 23.0 (39.0) | 47.8 (35.4) | 72.8 (44.9) | 13.7 (34.0) | 39.9 (70.8) | 67.9 (68.0) | 48.6 (21.8) | 48.0 (24.4) | 44.1 (36.5) | 70.8 (NA) — Only 1 subject so value cannot be calculated.

6. Secondary Outcome: Tmax of AT-007
Description: Time to reach maximum (peak) plasma drug concentration
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Groups:
- Part A Cohort 1: AT-007 0.5mg/kg; Part A Cohort 2: AT-007 5mg/kg; Part A Cohort 3: AT-007 10mg/kg; Part A Cohort 4: AT-007 20mg/kg; Part A Cohort 5: AT-007 40mg/kg: Following a single dose of AT-007 to Healthy Adult Subjects, sequential sampling was performed and Tmax calculated.
- Part B & C Cohort 1: AT-007 5mg/kg; Part B & C Cohort 2: AT-007 10mg/kg; Part B & C Cohort 3: AT-007 20mg/kg; Part B & C Cohort 4: AT-007 40mg/kg: Following multiple QD dose administration of AT-007 for 7 days in Healthy Adult Subjects, Tmax was calculated.
- Part D Cohort 1: AT-007 5mg/kg; Part D Cohort 2: AT-007 20mg/kg; Part D Cohort 3: AT-007 40mg/kg; Part D Extension Cohort 1: AT-007 20mg/kg DAY 30; Part D Extension Cohort 1: AT-007 20mg/kg DAY 60; Part D Extension Cohort 1: AT-007 20mg/kg DAY 90; Part D Extension Cohort 2: AT-007 40mg/kg DAY 30: Following multiple QD dose administration of AT-007 in Adults with Classic Galactosemia, Tmax was calculated.
Arm/Group | Part A Cohort 1: AT-007 0.5mg/kg | Part A Cohort 2: AT-007 5mg/kg | Part A Cohort 3: AT-007 10mg/kg | Part A Cohort 4: AT-007 20mg/kg | Part A Cohort 5: AT-007 40mg/kg | Part B & C Cohort 1: AT-007 5mg/kg | Part B & C Cohort 2: AT-007 10mg/kg | Part B & C Cohort 3: AT-007 20mg/kg | Part B & C Cohort 4: AT-007 40mg/kg | Part D Cohort 1: AT-007 5mg/kg | Part D Cohort 2: AT-007 20mg/kg | Part D Cohort 3: AT-007 40mg/kg | Part D Extension Cohort 1: AT-007 20mg/kg DAY 30 | Part D Extension Cohort 1: AT-007 20mg/kg DAY 60 | Part D Extension Cohort 1: AT-007 20mg/kg DAY 90 | Part D Extension Cohort 2: AT-007 40mg/kg DAY 30
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 9 | 7 | 4 | 4 | 4 | 9 | 8 | 6 | 1
hours | 4.00 [4.00 to 6.02] | 4.00 [2.00 to 4.00] | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 24.1] | 4.00 [4.00 to 8.00] | 4.00 [4.00 to 8.00] | 3.96 [2.00 to 8.00] | 4.00 [4.00 to 8.00] | 4.00 [4.00 to 6.07] | 4.00 [2.00 to 6.00] | 4.96 [4.00 to 8.00] | 4.00 [1.92 to 8.00] | 4.03 [1.97 to 8.02] | 4.01 [2.00 to 7.97] | 4.00 [2.00 to 4.33] | 4.17 [4.17 to 4.17]

7. Secondary Outcome: t1/2 of AT-007
Description: Terminal elimination half life
Time Frame: Part A: Sequential sampling at predose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 36, and 48 hours. Parts B, C, D: Determined using Day of Last Dose for the respective Part; predose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 36, and 48 hours.
Population: For Part D Extension, t1/2 was not performed so these cohorts are not presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Groups:
- Part A Cohort 1: AT-007 0.5mg/kg; Part A Cohort 2: AT-007 5mg/kg; Part A Cohort 3: AT-007 10mg/kg; Part A Cohort 4: AT-007 20mg/kg; Part A Cohort 5: AT-007 40mg/kg: Following a single dose of AT-007 to Healthy Adult Subjects, sequential sampling was performed and t1/2 calculated.
- Part B & C Cohort 1: AT-007 5mg/kg; Part B & C Cohort 2: AT-007 10mg/kg; Part B & C Cohort 3: AT-007 20mg/kg; Part B & C Cohort 4: AT-007 40mg/kg: Following multiple QD dose administration of AT-007 for 7 days in Healthy Adult Subjects, t1/2 was calculated.
- Part D Cohort 1: AT-007 5mg/kg; Part D Cohort 2: AT-007 20mg/kg; Part D Cohort 3: AT-007 40mg/kg: Following multiple QD dose administration of AT-007 in Adults with Classic Galactosemia, t1/2 was calculated.
Arm/Group | Part A Cohort 1: AT-007 0.5mg/kg | Part A Cohort 2: AT-007 5mg/kg | Part A Cohort 3: AT-007 10mg/kg | Part A Cohort 4: AT-007 20mg/kg | Part A Cohort 5: AT-007 40mg/kg | Part B & C Cohort 1: AT-007 5mg/kg | Part B & C Cohort 2: AT-007 10mg/kg | Part B & C Cohort 3: AT-007 20mg/kg | Part B & C Cohort 4: AT-007 40mg/kg | Part D Cohort 1: AT-007 5mg/kg | Part D Cohort 2: AT-007 20mg/kg | Part D Cohort 3: AT-007 40mg/kg
Number analyzed (Participants) | 6 | 4 | 6 | 1 | 2 | 6 | 8 | 9 | 7 | 3 | 3 | 4
hours | 13.7 (45.3) | 22.0 (92.6) | 10.3 (31.7) | 8.42 (NA) — Only 1 subject data available so cannot calculate. | 8.2 (7.55) | 13.1 (39.5) | 15.7 (79.9) | 9.76 (22.4) | 9.96 (27.4) | 13.9 (11.0) | 16.8 (56.6) | 16.1 (21.1)

8. Secondary Outcome: AUClast of AT-007
Description: Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration
Time Frame: Part A: Sequential sampling at predose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 36, and 48 hours. Parts B, C, D: Determined using Day of Last Dose for the respective Part at predose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 36, and 48 hours.
Population: For Part D Extension, AUClast was not performed so these cohorts are not presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour/mL
Groups:
- Part A Cohort 1: AT-007 0.5mg/kg; Part A Cohort 2: AT-007 5mg/kg; Part A Cohort 3: AT-007 10mg/kg; Part A Cohort 4: AT-007 20mg/kg; Part A Cohort 5: AT-007 40mg/kg: Following a single dose of AT-007 to Healthy Adult Subjects, sequential sampling was performed and AUClast calculated.
- Part B & C Cohort 1: AT-007 5mg/kg; Part B & C Cohort 2: AT-007 10mg/kg; Part B & C Cohort 3: AT-007 20mg/kg; Part B & C Cohort 4: AT-007 40mg/kg: Following multiple QD dose administration of AT-007 for 7 days in Healthy Adult Subjects, AUClast was calculated.
- Part D Cohort 1: AT-007 5mg/kg; Part D Cohort 2: AT-007 20mg/kg; Part D Cohort 3: AT-007 40mg/kg: Following multiple QD dose administration of AT-007 in Adults with Classic Galactosemia, AUClast was calculated.
Arm/Group | Part A Cohort 1: AT-007 0.5mg/kg | Part A Cohort 2: AT-007 5mg/kg | Part A Cohort 3: AT-007 10mg/kg | Part A Cohort 4: AT-007 20mg/kg | Part A Cohort 5: AT-007 40mg/kg | Part B & C Cohort 1: AT-007 5mg/kg | Part B & C Cohort 2: AT-007 10mg/kg | Part B & C Cohort 3: AT-007 20mg/kg | Part B & C Cohort 4: AT-007 40mg/kg | Part D Cohort 1: AT-007 5mg/kg | Part D Cohort 2: AT-007 20mg/kg | Part D Cohort 3: AT-007 40mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 9 | 7 | 4 | 4 | 4
microgram*hour/mL | 12.6 (44.7) | 89.0 (18.5) | 158 (35.0) | 352 (75.0) | 624 (28.0) | 181 (44.3) | 311 (47.4) | 592 (26.9) | 1110 (50.2) | 172 (25.3) | 698 (21.8) | 1006 (62.3)

9. Secondary Outcome: AUCinf of AT-007
Description: Area under the plasma concentration-time curve from time zero extrapolated to infinity
Time Frame: Part A: Sequential sampling at predose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 36, and 48 hours. Part D: Determined using Day 1 with sampling at predose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 36, and 48 hours.
Population: AUCinf was only calculated for all cohorts of Part A and on Day 1 of Part D. It was not calculated for Parts B, C, or D Extension so those cohorts are not presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour/mL
Groups:
- Part A Cohort 1: AT-007 0.5mg/kg; Part A Cohort 2: AT-007 5mg/kg; Part A Cohort 3: AT-007 10mg/kg; Part A Cohort 4: AT-007 20mg/kg; Part A Cohort 5: AT-007 40mg/kg: Following a single dose of AT-007 to healthy subjects, AUCinf was calculated.
- Part D Cohort 1: AT-007 5mg/kg; Part D Cohort 2: AT-007 20mg/kg; Part D Cohort 3: AT-007 40mg/kg: Following the first dose of AT-007 to adult subjects with Classic Galactosemia, AUCinf was calculated.
Arm/Group | Part A Cohort 1: AT-007 0.5mg/kg | Part A Cohort 2: AT-007 5mg/kg | Part A Cohort 3: AT-007 10mg/kg | Part A Cohort 4: AT-007 20mg/kg | Part A Cohort 5: AT-007 40mg/kg | Part D Cohort 1: AT-007 5mg/kg | Part D Cohort 2: AT-007 20mg/kg | Part D Cohort 3: AT-007 40mg/kg
Number analyzed (Participants) | 5 | 2 | 6 | 1 | 2 | 4 | 3 | 3
microgram*hour/mL | 14.3 (43.7) | 81.8 (15.1) | 169 (35.3) | 163 (NA) — Only 1 subject had data available so cannot calculate this. | 655 (0.45) | 109 (28.2) | 518 (65.2) | 1327 (17.2)

10. Secondary Outcome: Maximal Galactitol Reduction in Plasma
Description: Disease-Specific Biomarker in Classic Galactosemia Patients
Time Frame: Part D: Samples at predose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 36, and 48 hours on days 1, 12, 32. Part D Extension: Samples at predose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 36, and 48 hours on days 1, 30, 60, & 90.
Population: Part D Extension Cohort 2 40mg/kg ended early at Day 30 as recommended by Monitoring Committee. As such, there are no results for this outcome measure for the Part D Extension Cohort 2 40mg/kg.
Measure: Mean (Standard Deviation); unit: maximal change from baseline in ng/mL
Groups:
- Part D Cohort 1: AT-007 5mg/kg; Part D Cohort 2: AT-007 20mg/kg; Part D Cohort 3: AT-007 40mg/kg: Adults with Classic Galactosemia had galactitol plasma levels assessed predose after 32 days of AT-007 administration
- Part D Placebo Comparator: Adults with Classic Galactosemia had galactitol plasma levels assessed predose after 32 days of matched placebo administration
- Part D Extension AT-007 20mg/kg: Adults with Classic Galactosemia had galactitol plasma levels assessed predose after 30, 60, and 90 days of AT-007 administration. Maximal reduction of galactitol at any of the time points measured was calculated.
- Part D Extension Placebo Comparator: Adults with Classic Galactosemia had galactitol plasma levels assessed predose after 30, 60, and 90 days of matched placebo administration. Maximal reduction of galactitol at any of the time points measured was calculated.
Arm/Group | Part D Cohort 1: AT-007 5mg/kg | Part D Cohort 2: AT-007 20mg/kg | Part D Cohort 3: AT-007 40mg/kg | Part D Placebo Comparator | Part D Extension AT-007 20mg/kg | Part D Extension Placebo Comparator
Number analyzed (Participants) | 4 | 4 | 4 | 5 | 9 | 4
maximal change from baseline in ng/mL | -475 (305) | -1175 (239) | -1259 (220) | -393 (239) | -974.4 (322.42) | -344.0 (449.67)

11. Secondary Outcome: Galactose Concentration in Plasma
Description: Disease-Specific Biomarker in Classic Galactosemia Patients
Time Frame: Part D: Day 32. Part D Extension: Days 30, 60, & 90.
Population: Part D Extension Cohort 2 40mg/kg ended early at Day 30 as recommended by Monitoring Committee. As such, there are no results for this outcome measure for the Part D Extension Cohort 2 40mg/kg. Part D Extension Cohort 1 of AT-007 20mg/kg is presented for Days 30, 60, and 90.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Groups:
- Part D Cohort 1: AT-007 5mg/kg; Part D Cohort 2: AT-007 20mg/kg; Part D Cohort 3: AT-007 40mg/kg: Adults with Classic Galactosemia had galactose plasma levels assessed predose after 32 days of AT-007 administration
- Part D Placebo Comparator: Adults with Classic Galactosemia had galactose plasma levels assessed predose after 32 days of matched placebo administration
- Part D Extension AT-007 20mg/kg Day 30: Adults with Classic Galactosemia had galactose plasma levels assessed predose after 30 days of AT-007 administration.
- Part D Extension AT-007 20mg/kg Day 60: Adults with Classic Galactosemia had galactose plasma levels assessed predose after 60 days of AT-007 administration
- Part D Extension AT-007 20mg/kg Day 90: Adults with Classic Galactosemia had galactose plasma levels assessed predose after 90 days of AT-007 administration
- Part D Extension Placebo Comparator Day 30: Adults with Classic Galactosemia had galactose plasma levels assessed predose after 30 days of matched placebo administration
- Part D Extension Placebo Comparator Day 60: Adults with Classic Galactosemia had galactose plasma levels assessed predose after 60 days of matched placebo administration
- Part D Extension Placebo Comparator: Adults with Classic Galactosemia had galactose plasma levels assessed predose after 90 days of matched placebo administration
Arm/Group | Part D Cohort 1: AT-007 5mg/kg | Part D Cohort 2: AT-007 20mg/kg | Part D Cohort 3: AT-007 40mg/kg | Part D Placebo Comparator | Part D Extension AT-007 20mg/kg Day 30 | Part D Extension AT-007 20mg/kg Day 60 | Part D Extension AT-007 20mg/kg Day 90 | Part D Extension Placebo Comparator Day 30 | Part D Extension Placebo Comparator Day 60 | Part D Extension Placebo Comparator
Number analyzed (Participants) | 4 | 4 | 4 | 5 | 9 | 7 | 6 | 4 | 3 | 3
percent change from baseline | 8.94 (8.71) | -27.8 (29.3) | 25.4 (69.5) | 39.8 (62.7) | -153.78 (381.475) | 52.29 (170.753) | 30.42 (102.15) | 139.75 (273.418) | 98.67 (132.115) | 130.00 (101.059)

12. Secondary Outcome: Galactose-1-Phosphate (Gal-1p) Concentration in Plasma
Description: Disease-Specific Biomarker in Classic Galactosemia Patients
Time Frame: Part D: Day 32. Part D Extension: Days 30, 60, & 90.
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percent change from baseline
Groups:
- Part D Cohort 1: AT-007 5mg/kg; Part D Cohort 2: AT-007 20mg/kg; Part D Cohort 3: AT-007 40mg/kg: Adults with Classic Galactosemia had gal-1p plasma levels assessed predose after 32 days of AT-007 administration
- Part D Placebo Comparator: Adults with Classic Galactosemia had gal-1p plasma levels assessed predose after 32 days of matched placebo administration
- Part D Extension AT-007 20mg/kg Day 30: Adults with Classic Galactosemia had gal-1p plasma levels assessed predose after 30 days of AT-007 administration.
- Part D Extension AT-007 20mg/kg Day 60: Adults with Classic Galactosemia had gal-1p plasma levels assessed predose after 60 days of AT-007 administration
- Part D Extension AT-007 20mg/kg Day 90: Adults with Classic Galactosemia had gal-1p plasma levels assessed predose after 90 days of AT-007 administration
- Part D Extension Placebo Comparator Day 30: Adults with Classic Galactosemia had gal-1p plasma levels assessed predose after 30 days of matched placebo administration
- Part D Extension Placebo Comparator Day 60: Adults with Classic Galactosemia had gal-1p plasma levels assessed predose after 60 days of matched placebo administration
- Part D Extension Placebo Comparator: Adults with Classic Galactosemia had gal-1p plasma levels assessed predose after 90 days of matched placebo administration
Arm/Group | Part D Cohort 1: AT-007 5mg/kg | Part D Cohort 2: AT-007 20mg/kg | Part D Cohort 3: AT-007 40mg/kg | Part D Placebo Comparator | Part D Extension AT-007 20mg/kg Day 30 | Part D Extension AT-007 20mg/kg Day 60 | Part D Extension AT-007 20mg/kg Day 90 | Part D Extension Placebo Comparator Day 30 | Part D Extension Placebo Comparator Day 60 | Part D Extension Placebo Comparator
Number analyzed (Participants) | 4 | 4 | 4 | 5 | 9 | 7 | 6 | 4 | 3 | 3
percent change from baseline | 5.71 (15.7) | 31.5 (6.78) | 7.86 (21.0) | 25.2 (8.74) | 33.1 (51.123) | 16.04 (43.218) | 4.87 (24.917) | 8.63 (24.473) | 14.03 (13.181) | 11.97 (21.511)

ADVERSE EVENTS:
Time Frame: Part A: 1 day; Part B&C: 7 days; Part D: 32 days; Part D Extension: 90 days
Groups:
- Part A Cohort 1: AT-007 0.5mg/kg; Part A Cohort 2: AT-007 5mg/kg; Part A Cohort 3: AT-007 10mg/kg; Part A Cohort 4: AT-007 20mg/kg; Part A Cohort 5: 40mg/kg: Single ascending doses of orally administered AT-007 were administered to healthy adult subjects.
- Part A Placebo Comparator: Single ascending doses of orally administered matched placebo were administered to healthy adult subjects.
- Part B & C Cohort 1: AT-007 5mg/kg; Part B & C Cohort 2: AT-007 10mg/kg; Part B & C Cohort 3: AT-007 20mg/kg; Part B & C Cohort 4: AT-007 40mg/kg: Multiple doses of orally administered AT-007 were administered to healthy adult subjects.
- Part B & C Placebo Comparator: Multiple doses of orally administered matched placebo were administered to healthy adult subjects.
- Part D Cohort 1: AT-007 5mg/kg; Part D Cohort 2: AT-007 20mg/kg; Part D Cohort 3: AT-007 40mg/kg; Part D Extension Cohort 1: 20mg/kg; Part D Extension Cohort 2: 40mg/kg: Multiple doses of orally administered AT-007 were administered to adult subjects with Classic Galactosemia.
- Part D Placebo Comparator; Part D Extension Placebo Comparator: Multiple doses of orally administered matched placebo were administered to adult subjects with Classic Galactosemia.
Arm/Group | Part A Cohort 1: AT-007 0.5mg/kg | Part A Cohort 2: AT-007 5mg/kg | Part A Cohort 3: AT-007 10mg/kg | Part A Cohort 4: AT-007 20mg/kg | Part A Cohort 5: 40mg/kg | Part A Placebo Comparator | Part B & C Cohort 1: AT-007 5mg/kg | Part B & C Cohort 2: AT-007 10mg/kg | Part B & C Cohort 3: AT-007 20mg/kg | Part B & C Cohort 4: AT-007 40mg/kg | Part B & C Placebo Comparator | Part D Cohort 1: AT-007 5mg/kg | Part D Cohort 2: AT-007 20mg/kg | Part D Cohort 3: AT-007 40mg/kg | Part D Placebo Comparator | Part D Extension Cohort 1: 20mg/kg | Part D Extension Cohort 2: 40mg/kg | Part D Extension Placebo Comparator
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10 | 0/6 | 0/8 | 0/10 | 0/9 | 0/8 | 0/4 | 0/4 | 0/4 | 0/6 | 0/9 | 0/2 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10 | 0/6 | 0/8 | 0/10 | 0/9 | 0/8 | 0/4 | 0/4 | 0/4 | 0/6 | 1/9 | 0/2 | 0/4
Other Adverse Events (participants affected / at risk) | 1/6 | 0/6 | 0/6 | 2/6 | 1/6 | 2/10 | 1/6 | 2/8 | 3/10 | 1/9 | 2/8 | 3/4 | 1/4 | 2/4 | 2/6 | 7/9 | 1/2 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A Cohort 1: AT-007 0.5mg/kg (N=6) | Part A Cohort 2: AT-007 5mg/kg (N=6) | Part A Cohort 3: AT-007 10mg/kg (N=6) | Part A Cohort 4: AT-007 20mg/kg (N=6) | Part A Cohort 5: 40mg/kg (N=6) | Part A Placebo Comparator (N=10) | Part B & C Cohort 1: AT-007 5mg/kg (N=6) | Part B & C Cohort 2: AT-007 10mg/kg (N=8) | Part B & C Cohort 3: AT-007 20mg/kg (N=10) | Part B & C Cohort 4: AT-007 40mg/kg (N=9) | Part B & C Placebo Comparator (N=8) | Part D Cohort 1: AT-007 5mg/kg (N=4) | Part D Cohort 2: AT-007 20mg/kg (N=4) | Part D Cohort 3: AT-007 40mg/kg (N=4) | Part D Placebo Comparator (N=6) | Part D Extension Cohort 1: 20mg/kg (N=9) | Part D Extension Cohort 2: 40mg/kg (N=2) | Part D Extension Placebo Comparator (N=4)
Liver Injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — There was 1 severe SAE of liver injury in 1 subject (20 mg/kg dosing) that was considered not related to study drug by the independent Liver Safety Adjudication Committee.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A Cohort 1: AT-007 0.5mg/kg (N=6) | Part A Cohort 2: AT-007 5mg/kg (N=6) | Part A Cohort 3: AT-007 10mg/kg (N=6) | Part A Cohort 4: AT-007 20mg/kg (N=6) | Part A Cohort 5: 40mg/kg (N=6) | Part A Placebo Comparator (N=10) | Part B & C Cohort 1: AT-007 5mg/kg (N=6) | Part B & C Cohort 2: AT-007 10mg/kg (N=8) | Part B & C Cohort 3: AT-007 20mg/kg (N=10) | Part B & C Cohort 4: AT-007 40mg/kg (N=9) | Part B & C Placebo Comparator (N=8) | Part D Cohort 1: AT-007 5mg/kg (N=4) | Part D Cohort 2: AT-007 20mg/kg (N=4) | Part D Cohort 3: AT-007 40mg/kg (N=4) | Part D Placebo Comparator (N=6) | Part D Extension Cohort 1: 20mg/kg (N=9) | Part D Extension Cohort 2: 40mg/kg (N=2) | Part D Extension Placebo Comparator (N=4)
Gastrointestinal Disorders (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
ALT Increased (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Infections/Infestations (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Musculoskelatal & Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nervous System (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Investigations (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General Disorders (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Seasonal Allergies (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Reproductive System Disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-09-03): https://cdn.clinicaltrials.gov/large-docs/11/NCT04117711/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-20): https://cdn.clinicaltrials.gov/large-docs/11/NCT04117711/SAP_001.pdf